CLINICAL TRIAL: NCT05926141
Title: Advanced Cooking Education (ACE) 4-H After School Club Pilot Study
Brief Title: Advanced Cooking Education Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0145840
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Adolescent Behavior; Nutrition, Healthy
Keywords: Adolescents; Nutrition intervention; Culinary programs
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: All participants enter a control phase for 12 weeks where they receive no intervention. After 12 weeks, the same group of participants receive the ACE intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control phase (No Intervention): After the first data collection session, participants spend 12 weeks and enter a "control phase" where they receive no intervention. At the end of the 12 weeks, participants will attend another data collection session.
- ACE intervention (Experimental): The ACE Program is a culturally inclusive, 4-H after school club where youth meet once a week for 12 weeks after school in person. They also receive groceries to make a meal 1 day a week.
  Interventions: Behavioral: ACE intervention

INTERVENTIONS:
Behavioral: ACE intervention — Participants attend the ACE Program for 12 weeks after school. On one assigned day of the week, participants attend ACE in person after school. The session begins with mindfulness exercises (15 minutes), professional development session (50 minutes), nutrition education lesson (20 minutes), and reflection period to talk about their experience in cooking lessons (25 minutes). On any day during the week, the students will make a dish using groceries they received (1 hour).
  Arms: ACE intervention

SUMMARY:
The aim of this study is to assess the impact of an in-person multi-component Advanced Cooking Education (ACE) 4-H after school program. The ACE Program consists of mindfulness, nutrition education, cooking labs, and professional development activities.

DETAILED DESCRIPTION:
The ACE program is conducted with 7th and 8th grade students attending New York City (NYC) Title I middle schools. Participants attend weekly sessions (2hour) after school to participate in mindfulness, nutrition lessons, and professional development activities. On another day in the week, students participate in cooking labs at their own time at their homes. The investigators hypothesize that after the program, adolescents' diet quality, cooking-related skills, stress levels will be improved compared to prior of the program.

ELIGIBILITY:
Inclusion Criteria:

* 7th and 8th grade students attending Title I funded schools in New York City
* Caregivers of the 7th and 8th grade students attending Title I funded schools in New York City

Exclusion Criteria:

* Do not speak/understand English
* Those who have previously participated in the Virtual ACE program (Feasibility Study)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Difference in change in diet quality between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Healthy Index Eating scores are calculated from three 24-hour diet records, range from 0-100. Higher score reflects higher alignment between one's diet and recommendations from Dietary Guidelines for Americans

SECONDARY OUTCOMES:
Difference in change in body mass index between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Height will be measured using stadiometer to nearest decimal point in cm. Weight is measured using scale to nearest decimal in kg. Body mass index calculated using kg/m^2.
Difference in change in body fat percentage between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Measured using a scale to nearest decimal
Difference in change in waist circumference between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Measured using a waist circumference tape to the nearest decimal in cm
Difference in change in dermal carotenoids level between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Measured using the Veggie Meter device, range from 0-800. Higher score acts as proxy for increased fruits and vegetables consumption
Difference in change in household food security between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Short form food security survey module by the USDA. Higher scores indicate lower food security status. Min=0, Max=6
Difference in change in culinary skills between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  iCook program youth culinary skill survey with 5-point likert scale questions with higher scores indicate higher skill level (better outcome). Min=7, Max=35
Difference in change in culinary self-efficacy between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  iCook program youth culinary self-efficacy survey with 5-point likert scale questions with higher scores indicate higher skill level (better outcome). Min=6, Max=30
Difference in change in culinary attitudes between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Cooking with kids survey with 5-point likert scale questions with higher scores indicate more positive attitude (better outcome). Min=6, Max=30
Difference in change in perceived stress between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Used the Cohen perceived stress scale. Higher scores mean increased stress (worse outcome). Min=0, Max=40
Difference in change in food neophobia between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  FNTT10 survey with 5-point likert scale questions, higher scores mean less neophobia (better outcome). Min=10, Max=50.
Difference in change in sense of purpose between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Used the Clarement Purpose Scale survey questions, higher scores mean higher sense of purpose (better outcome). Min=12, Max=60
Difference in change in social and emotional competency between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Used the SEC survey by CASEL, higher scores mean higher competence (better outcome). Min=17, Max= 68
Difference in change in family mealtime beliefs between intervention phase (12-24wk) and control phase (0wk-12wk) | 0 weeks, 12 weeks, 24 weeks, 48 weeks
  Calculated based on the Fulkerson family mealtime survey. A total of 9 questions that are scored independently. Each: Min=1, Max=4. Higher scores indicate better family mealtime practices (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Tashara M Leak, PhD RD, Principal Investigator — Cornell University
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No